CLINICAL TRIAL: NCT05558306
Title: Association Between Radiographic and Clinical Outcome in Distal Radius Fractures: A Prospective Cohort Study With a 1-year Follow-up in 368 Patients
Brief Title: Radiological vs Clinical Outcome in DRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS_DRF_Outcome
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment protocol (Other): All patients were treated according to the treatment protocol with cast for minimally displaced fractures and surgery for displaced fractures.
  Interventions: Procedure: Surgery of distal radius fracture; Procedure: Reduction and cast treatment of distal radius fracture

INTERVENTIONS:
Procedure: Surgery of distal radius fracture — Surgery of distal radius fracture for displaced fractures
Procedure: Reduction and cast treatment of distal radius fracture — Reduction and cast treatment of distal radius fracture for minimally displaced fractures

SUMMARY:
Background: Several studies have investigated the degree of final displacement and its association with clinical outcome. There is still no consensus on the importance of radiological outcome and published studies do not use the same criteria for an acceptable alignment. Previous reports have used a linear or a dichotomized exposure in the statistical analysis, but no study has investigated a nonlinear association.

Methods: We included 438 patients treated for a distal radius fracture (DRF) with either reduction and cast immobilization or surgery. Radiographic outcomes were determined by radiographs 3 months after the injury. Clinical outcome was determined by QuickDASH (qDASH), ROM and grip strength at 1-year after the injury. Nonlinear correlations were analysed with cubic splines.

ELIGIBILITY:
Inclusion Criteria:

- Patients with distal radius fracture between 15 and 74 years, with closed physes of the distal radius and ulna.

Exclusion Criteria:

* Dementia
* Previous fracture to the ipsilateral wrist
* Open fracture
* Other concomitant or existing damage or injury to the wrist
* Galeazzi fracture
* Rheumatoid arthritis
* Alcohol or drug abuse
* Neurologic impairment

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
quickDASH | 12 months
  The DASH is a 30-item PROM questionnaire that evaluates the upper extremity [115]. The qDASH is a shortened version with 11 questions that can be used instead of the full 30-item questionnaire [114]. Both are validated for use in upper extremity disorders [114,115]. Neither is specific for wrist function and both yield scores from 0 to 100, where lower scores indicate a better outcome.
Range of motion | 12 months
  The active ROM of the radiocarpal joint and the radioulnar joints were measured in both hands using a standard goniometer. The arcs of flexion-extension, pronation-supination and radial-ulnar deviation were recorded. Total ROM was calculated as the sum of these three arcs. The loss of ROM in the fractured wrist was expressed in angular degrees compared to the contralateral uninjured wrist [126].
  Independent occupational therapists, blinded to the radiological outcome, measured objective function, including grip strength and active ROM.
Grip strength | 12 months
  Grip strength was measured in a sitting position with the elbow in 90° of flexion, neutral rotation and wrist 0°-30° extension using a JAMAR dynamometer [122]. To prevent it from falling, the examiner may support the JAMAR dynamometer. Both hands are examined, starting with the uninjured hand. Three strength tests were conducted during the assessment of grip strength, with the mean score of the three tests recorded for analysis. Grip strength was adjusted by 10% for the non-dominant hand [123]. The contralateral wrist was used as an internal control. Grip strength was expressed as a percentage (the ratio to the uninjured wrist) and the absolute loss in kilograms comparing the fractured wrist to the uninjured wrist.
  Independent occupational therapists, blinded to the radiological outcome, measured objective function, including grip strength and active ROM.

REFERENCES:
- [Derived] Schmidt V, Gordon M, Tagil M, Sayed-Noor A, Mukka S, Wadsten M. Association Between Radiographic and Clinical Outcomes Following Distal Radial Fractures: A Prospective Cohort Study with 1-Year Follow-up in 366 Patients. J Bone Joint Surg Am. 2023 Aug 2;105(15):1156-1167. doi: 10.2106/JBJS.22.01096. Epub 2023 May 12. PMID 37172109